CLINICAL TRIAL: NCT00496847
Title: Study on the Efficacy and Safety of PERIOGEN in the Treatment of Periodontal Bone Defect - A Double-blind, Controlled, Randomised,Parallel,Multi-centre Study
Brief Title: Efficacy and Safety of PERIOGEN in the Treatment of Periodontal Bone Defect
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virchow Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VB023/07
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2009-11

CONDITIONS: Intrabony Periodontal Defect
Keywords: rhPDGF,; periodontal disease
MeSH Terms: conditions — Periodontal Diseases | interventions — beta-tricalcium phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug Group (Experimental): PERIOGEN
  Interventions: Drug: PERIOGEN
- Control group (Active Comparator): Beta TCP alone
  Interventions: Drug: Beta TCP alone

INTERVENTIONS:
Drug: PERIOGEN — Implantation of rhPDGF-BB (0.3 mg/ml) + β-TCP (0.5 g)
  Arms: Drug Group
Drug: Beta TCP alone — Implantation of β-TCP (0.5 g) alone
  Arms: Control group

SUMMARY:
PERIOGEN, containing rhPDGF and -beta-TCP, promotes gingival healing and corrects periodontal defects. This study will test the safety and efficacy of PERIOGEN in the treatment of periodontal disease

DETAILED DESCRIPTION:
Sixty eligible patients with periodontal defect will randomly receive either beta-TCP implantation (control group) or PERIOGEN implantation, containing beta-TCP and rhPDGF (drug group). The specified primary and secondary end points related to efficacy and safety will be assessed during 6 months study period.

ELIGIBILITY:
Inclusion Criteria:

1. Probing depth ≥7 mm at baseline
2. Presence of ≥4 mm vertical bone defect with at least 1 bony wall after surgical debridement.
3. Adequate keratinized tissue to permit complete tissue coverage of defect.
4. Radiographic base of defect ≥3 mm coronal to the apex of the tooth.

Exclusion Criteria:

1. Failure to maintain adequate oral hygiene (plaque index>2)
2. Pregnant and lactating women
3. History of oral cancer or HIV
4. Periodontal surgery on treatment-targeted tooth within the last year.
5. Tooth mobility greater than grade II.
6. Study tooth exhibiting a class III furacation defect
7. Localized aggressive periodontitis
8. Radiographic signs of untreated acute infection at the surgical site
9. Recent history of smoking more than 20 cigarettes/day
10. Known allergy to E.coli-derived products
11. Using an investigational therapy within the past 30 days.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
1.Area under curve (AUC) of clinical attachment level (CAL) gain (0-24 weeks) 2.Extent of linear bone growth (LBG) and percentage of bone fill (%BF) at 6 months. | 6 months

SECONDARY OUTCOMES:
1.Changes in CAL gain, probing depth and gingival recession at 3 and 6 months. 2.Incidence of adverse events. | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: A Jayakumar, MDS, Principal Investigator — Sri Sai Dental college of surgery, Vikarabad, RR Dist, AP, India.
Locations (1):
- Sri Sai Dental college of surgery, Vikarabad,, RR Dist, Andhra Pradesh, India

REFERENCES:
- [Derived] Jayakumar A, Rajababu P, Rohini S, Butchibabu K, Naveen A, Reddy PK, Vidyasagar S, Satyanarayana D, Pavan Kumar S. Multi-centre, randomized clinical trial on the efficacy and safety of recombinant human platelet-derived growth factor with beta-tricalcium phosphate in human intra-osseous periodontal defects. J Clin Periodontol. 2011 Feb;38(2):163-72. doi: 10.1111/j.1600-051X.2010.01639.x. Epub 2010 Dec 6. PMID 21133980